CLINICAL TRIAL: NCT00458094
Title: Activating Consumers to Exercise in Community Psychiatry Through Peer Support
Brief Title: Peer Support for Increasing Physical Activity in People With Serious Mental Illnesses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH078613 (NIH); R34MH078613 (NIH); DAHBR 96-BHB
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Schizophrenia; Depression; Bipolar Disorder; Anxiety Disorders; Cognitive Disorders; Personality Disorders
Keywords: Exercise; Mental Illness; Community Psychiatry; Peer Support; Mental Disorders
MeSH Terms: conditions — Schizophrenia; Depression; Bipolar Disorder; Anxiety Disorders; Cognitive Dysfunction; Personality Disorders; Motor Activity; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive the peer-supported physical activity intervention
  Interventions: Behavioral: Physical activity intervention with peer support (PA+PS)
- 2 (Active Comparator): Participants will receive physical activity without peer support
  Interventions: Behavioral: Physical activity intervention without peer support (PA)

INTERVENTIONS:
Behavioral: Physical activity intervention with peer support (PA+PS) — Participants in the PA+PS group will have three exercise sessions each week for 4 months, which will include group exercise classes and open gym hours for supervised individual exercise. They will also meet with a peer educator once a week for 15 minutes. Peer educators will provide emotional, informational, instrumental, and appraisal support that is aimed to motivate participants to partake in the exercise sessions.
  Arms: 1
Behavioral: Physical activity intervention without peer support (PA) — Participants in the PA group will attend the three weekly exercise sessions for 4 months but will not attend meetings with the peer educator.
  Arms: 2

SUMMARY:
This study will determine the effectiveness of a peer support system in increasing physical activity and effecting health behavior change in people with serious mental illnesses.

DETAILED DESCRIPTION:
People with serious mental illnesses (SMIs) are, by definition, significantly functionally impaired by the illness for an indefinite period of time. Schizophrenia, major depression, and bipolar disorder are considered SMIs. Severe anxiety disorders, cognitive disorders, and some personality disorders are sometimes categorized as SMIs, as well. The rate of obesity among people with SMIs is higher than that of people without mental illnesses. This disparity may be due to the negative symptoms that people with SMIs experience, such as vulnerability to stress, extreme dependency, and lack of motivation. This study will design and test a culturally appropriate physical activity intervention based on a peer support model for people with SMIs in an urban community psychiatry program. The intervention will be evaluated to determine its effectiveness in increasing physical activity and effecting health behavior change in people with SMIs.

Participants in this 4-month, open-label study will be randomly assigned to participate in either a physical activity intervention with peer support (PA+PS) or a physical activity intervention without peer support (PA). Participants in the PA+PS group will have three exercise sessions each week, which will include group exercise classes and open gym hours for supervised individual exercise. They will also meet with a peer educator once a week for 15 minutes. Peer educators will provide emotional, informational, instrumental, and appraisal support that is aimed to motivate participants to partake in the exercise sessions. Participants in the PA group will attend the three weekly exercise sessions but will not attend meetings with the peer educator. All outcomes will be assessed at a follow-up visit at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the Johns Hopkins Community Psychiatry program
* Plans to remain in Baltimore for 8 months after study entry
* If currently breastfeeding, has received approval from a physician to participate in the study

Exclusion Criteria:

* Any condition that would make weight loss medically inadvisable
* Diagnosis of or treatment for cancer (except non-melanoma skin cancer) within 2 years prior to study entry
* Liver failure
* History of anorexia nervosa
* Pregnant or planning to become pregnant during the study
* Inability to walk or participate in an exercise class
* Consumes more than 14 alcoholic drinks per week
* Symptoms of angina or a cardiovascular event within 6 months prior to study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Measured at Month 4

SECONDARY OUTCOMES:
Weight | Measured at Month 4
Waist circumference | Measured at Month 4
Physical activity | Measured at Month 4
Health status | Measured at Month 4
Center for Epidemiology Depression Scale | Measured at Month 4
Exercise-related self-efficacy | Measured at Month 4
General perceived efficacy | Measured at Month 4
Participation | Measured at Month 4

CONTACTS AND LOCATIONS:
Overall Officials: Gail L. Daumit, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States